CLINICAL TRIAL: NCT03677895
Title: What Factors Are Associated With Prognosis of Rotator Cuff Disorder After Subacromial Hyaluronic Acid Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02-006C
Record Dates: First submitted 2018-09-09; First posted 2018-09-19 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Rotator Cuff Impingement Syndrome
Keywords: rotator cuff disorder
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: patients with rotator cuff disorders receving subacromial hyaluronic acid injection
Masking Description: outcome assessor does not know the rotator cuff condition of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with rotator cuff disorders (Experimental): patients with rotator cuff disorders, including impingment, rotator cuff disorders and rotator cuff tear receiving hyaluronic acid injection over subacromial bursa
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Drug: Hyaluronic Acid — Hyaluronic Acid 2cc into subacromial bursa at weeks 0, 2 and 4
  Other Names: hyruan

SUMMARY:
To evaluate the correlations between structure of supraspinatus tendon (impingement, tendinopathy or partial tear, as well as full thickness tear) on ultrasonography and its response to subacromial hyaluronic acid injection in rotator cuff disease patients

DETAILED DESCRIPTION:
Objective: To evaluate the correlations between structure of supraspinatus tendon (impingement, tendinopathy or partial tear, as well as full thickness tear) on ultrasonography and its response to subacromial hyaluronic acid injection in rotator cuff disease patients and also investigate the factors associated with clinically important improvement after subdeltoid hyaluronic acid for rotator cuff disorder.

Design: Prospective, longitudinal comparison study.

Participants: Patients with rotator cuff disease

Intervention: Three subacromial injection with hyaluronic acid with 2 week-interval.

Main Outcome Measures: Visual analog scale (VAS) of the shoulder pain, Constant score, SPADI score, and angles of active shoulder range of motion (flexion, abduction, external rotation, and internal rotation) at pre-treatment, post-treatment at week 4 and post-treatment at week 12.

ELIGIBILITY:
Inclusion criteria were patients

1. with clinically and ultrasonographically diagnosed rotator cuff disease of the shoulder-impingement, tendinosis and tear;
2. who reported shoulder pain more than 3 months;

Exclusion Criteria:

1. presence of another medical or psychological condition, including cancer, rheumatoid arthritis, endocrine disease (i.e., diabetes), major depression, or schizophrenia;
2. previous major trauma history at currently affected shoulder; 3 primary osteoarthritis of the glenohumeral joint in a simple radiograph; 4previous injection history at the affected shoulder within 3 months

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
constant shoulder score | 12 weeks
  the total constant score ranges from 0 to 100 points, with higher scores indicative of better function. The score is divided into four sections: pain, activity of daily living, ROM and the total constant score ranges from 0 to 100 points, with higher scores indicative of better function. The score is divided into four sections: pain, activity of daily living, ROM and strength

SECONDARY OUTCOMES:
pain intensity measured by visual analog scale | 0, 6, 12 weeks
  pain intensity was measured by visual analog scale. the total score ranges from 0 to 10 points, with higher scores indicative of more painful
Shoulder Pain And disability index | 0, 6, 12 weeks
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
glenohumeral joint range of motion | 0, 6, 12 weeks
  Shoulder flexion, abduction, external rotation and internal rotation were measured with goniometer with patient in supine position

CONTACTS AND LOCATIONS:
Overall Officials: Jia Chi Wang, MD, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan